CLINICAL TRIAL: NCT03451435
Title: N-Acetyl Cysteine Helps Pulp Stem Cells Differentiate During Endodontic Revascularization
Brief Title: N-Acetyl Cysteine Protects Pulpal Stem Cells in Endodontic Revascularization
Acronym: NAC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David C. Han, DDS, MS, Research Scientist and Clinical Director, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-001024
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention will be administered in this group as it serves as a control group.
- NAC Treatment (Experimental): N-Acetyl Cysteine treatment during root canal revascularization
  Interventions: Drug: N acetyl cysteine

INTERVENTIONS:
Drug: N acetyl cysteine — N acetyl cysteine at 20mM will be utilized as the final stage of irrigation prior to induction of bleeding during endodontic revascularization procedure.
  Arms: NAC Treatment

SUMMARY:
Pulp re-vascularization/regeneration is a procedure performed to allow pulpal stem cells to survive and/or differentiate to allow immature tooth root structures to grow to full maturity. Currently, the procedure includes disinfection of the necrotic root canal space and induction of bleeding to potentiate pulpal stem cell differentiation to allow root growth on an immature root. A number of studies conducted previously demonstrate that N-acetyl cysteine (NAC) potentiates differentiation of pulpal stem/stromal cells and protects pulpal cells from apoptosis. 14-18 human subjects will be recruited forming two groups where pulp re-vascularization/regeneration procedures will be performed with or without the use of NAC treatment prior to induction of bleeding. Recall follow-up appointments will be done at 6 months and 1 year post treatment with subsequent yearly appointments until full root growth has been achieved.

DETAILED DESCRIPTION:
We will recruit 14-18 patients under the age of 18 by means of advertising at UCLA. Two groups will be formed, one with NAC treatment during endodontic revascularization and one without. Each patient will have an adult tooth where the following criteria are met:

* Tooth with necrotic pulp and immature apex(apices)
* Pulp space is not needed for post/core, final restoration
* Compliant patient who is willing to come for at least 2-3 treatment appointments and 2-3 follow-up recall appointments.
* Patients are not allergic to calcium hydroxide intra-canal medicament

Appropriate consent forms will be obtained by the patient and the patient's parent or legal guardian. If we recruit 18 patient, 9 patients will be under regenerative endodontic therapy/re-vascularization with NAC and 9 patients without NAC.

The following procedures will be applied to the patients.

First Appointment:

* Local anesthesia administration, dental dam isolation and access
* Copious, gentle irrigation with 20mL NaOCL (sodium hypochlorite) using an irrigation system that minimizes the possibility of extrusion of irrigants into the periapical spaces. The concentration of NaOCL will be low (1.5%, 20mL/canal for 5 minutes). Afterwards, irrigation with 17% EDTA (20mL/canal for 5 minutes) will be done. Irrigating needle position should be about 1mm from root end, to minimize cytotoxicity to stem cells in the apical tissues.
* Dry canals with paper points
* Place calcium hydroxide into canal(s) delivered via syringe
* Seal access with 3-4mm of a temporary restorative material such as CavitTM, IRMTM or glass ionomer. Dismiss patient for 2-4 weeks.

Second Appointment:

* Assess response to initial treatment. If there are signs/symptoms of persistent infection, consider repeating the procedures of the First appointment.
* Anesthesia with 3% mepivacaine without vasoconstrictor, dental dam isolation
* Copious gentle irrigation with 20mL of 17% EDTA
* Take a radiograph to ensure previous calcium hydroxide has been fully removed form the canal system
* Dry with paper points
* For study patients only: Irrigate canal system with NAC (20mM NAC, 30mL/canal) gently for 10 minutes and then dry canal(s) with paper points
* Create bleeding into the canal system by over-instrumenting (endo file, endo explorer). Induce bleeding by rotating a pre-curved (approximately 45 degrees at the apical 1-2mm of file) K-file at 2mm past the apical foramen with the goal of having the entire canal filled with blood to the level of the cemento-enamel junction.
* Stop the bleeding at a level that allows for 3-4mm of restorative material. Place a resorbable matrix (CollaPlugTM, CollacoteTM, CollatTapeTM) over the blood clot if necessary to achieve a better stop for mineral trioxide aggregate (MTA) or Bioceramic fast set putty (BC). Place white MTA as capping material on top of the resorbable matrix.
* The access is closed with 3-4mm layer of glass ionomer (Fuji IXTM, GC America, Alsip, IL), composite or alloy over the capping material. For resin modified glass ionomers and composite, 40 seconds of light curer will be done.

Follow-up recall appointments: Clinical and Radiographic exam

* Extra-oral examination: No pain, extra-oral swelling nor extra-oral sinus tract
* Intra-oral examination: No pain, intra-oral swelling of mucosa nor intra-oral sinus tract
* Take 1 straight on periapical radiograph and 1 angled periapical radiograph. Resolution of apical radiolucency (often observed within 6-12months).
* Record any increased width of root walls (this is generally observed before apparent increase in root length and often occurs 12-24 months after treatment)
* Record any increase in root length (in mm)
* Test vitality of pulp with Endo-Ice and Electric pulp tester (EPT).
* Record which goals have been attained (primary, secondary and/or tertiary)

The degree of success of RET is measured by the extent to which it is possible to attain primary, secondary and tertiary goals:

* Primary goal: The elimination of symptoms and the evidence of bony healing
* Secondary goal: Increased root wall thickness and/or increased root length
* Tertiary goal: Positive response to vitality testing

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include the following:

  1. Subjects will be self and parent-reported as healthy individuals with no significant medical issues.
  2. Radiographic assessment will determine that root(s) have not grown to completion

  2) Vitality tests (cold testing with Endo ice and Electric pulp testing) will determine the tooth to be necrotic 3) Palpation and percussion tests may or may not be positive 4) Probings will be within 1-5mm 5) Patient will commit to coming to 2-3 treatment appointments lasting 1-3 hours each. Thereafter, patient will commit to come for followup recall appointments 6 and 12 months following last treatment appointment.

  6) Patient must be able to tolerate sitting in a dental chair for 1-3 hours. 7) Patient will be in the age range of 6 to 18 years

Exclusion Criteria:

* Exclusion criteria include patients who cannot tolerate sitting in a dental chair due to anxiety for 1-2 hours.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change of Root length | 6 months and 1 year
  Change of root length in millimeters over time

CONTACTS AND LOCATIONS:
Overall Officials: David C Han, DDS, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles Dept of Graduate Endodontics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No